CLINICAL TRIAL: NCT02262715
Title: A Phase 1, Randomized, 3-way Crossover, Open-label Study to Assess the Drug-drug Interaction Between VX-787 and Tamiflu®, Followed by a Double-blind, Randomized, Placebo-controlled Study to Collect Safety, Tolerability and Pharmacokinetics of VX-787, in Healthy Subjects
Brief Title: A Study to Assess the Drug-Drug Interaction Between VX-787 and Oseltamivir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Infectious Diseases BVBA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR105145; VX-787FLZ1001 (Other: Janssen Infectious Diseases BVBA); 2014-002528-28 (EudraCT Number)
Record Dates: First submitted 2014-08-26; First posted 2014-10-13 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: Oseltamivir; VX-787
MeSH Terms: interventions — pimodivir; Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 (Experimental): Participants will receive in random order Treatment A (VX-787, 600 mg tablet 2 times a day on Day 1 to 4, followed by VX 787, 600 mg tablet on Day 5); Treatment B (Oseltamivir, 75 mg capsule 2 times a day on Day 1 to 4, followed by oseltamivir 75 mg capsule in the morning on Day 5) or Treatment C (VX-787, 600 mg tablet, 2 times a day orally + oseltamivir, 75 mg capsule, 2 times a day on Day 1 to 4, followed by a single dose of VX-787, 600 mg + oseltamivir, 75 mg capsule on Day 5). Each participant will receive all three treatments (Treatment A, B and C) in a random sequence.
  Interventions: Drug: VX-787; Drug: Oseltamivir
- Part 2 VX-787 (Experimental): Participants will receive VX-787, 600 mg, tablet 2 times a day, orally on Day 1 to Day 9, followed by single dose of VX-787, 600 mg on Day 10.
  Interventions: Drug: VX-787
- Part 2 Placebo (Experimental): Participants will receive placebo matching to VX-787, 2 times a day, orally on Day 1 to Day 9, followed by single dose of matching placebo on Day 10.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: VX-787 — Participants will receive VX-787, 600 mg either two times a day or once a day in either of the Part.
  Arms: Part 1; Part 2 VX-787
Drug: Oseltamivir — Participants will receive Oseltamivir 75 mg either two times a day or once a day in either of the Part.
  Arms: Part 1
Other: Placebo — Participants will receive placebo matching to VX-787 either two times a day or or once a day.
  Arms: Part 2 Placebo

SUMMARY:
The purpose of this study is to investigate the drug-drug interaction between VX-787 and oseltamivir, when co-administered at steady-state in healthy participants. In addition the safety, tolerability and pharmacokinetics (the study of the way a drug enters and leaves the blood and tissues over time) of VX-787 will be assessed.

DETAILED DESCRIPTION:
This study consists of 2 parts. Part 1 is an open-label (a medical research study in which participants and researchers are told which treatments the participants are receiving), randomized (treatment group assigned by chance), 3-way crossover (a method used to switch participants from one treatment group to another in a clinical trial) study to estimate drug-drug interaction between VX-787 and oseltamivir. It consists of 3 phases: a Screening phase, a Treatment phase and a Follow-up phase. Treatment phase will include 3 treatment sessions, each of the participant will receive Treatment A (VX-787, 600 milligram [mg] 2 times a day on Day 1 to 4, followed by a single dose of VX 787, 600 mg on Day 5); Treatment B (Oseltamivir, 75 mg 2 times a day on Day 1 to 4, followed by a single dose of oseltamivir 75 mg on Day 5) and Treatment C (VX-787, 600 mg 2 times a day + oseltamivir, 75 mg 2 times a day on Day 1 to 4, followed by a single dose of VX-787, 600 mg + a single dose of oseltamivir, 75 mg on Day 5). Each treatment session will be separated by a wash-out period of 5 days. The order each participant will receive treatments A, B and C will be decided at randomization.

Part 2 is double-blind (a medical research study in which neither the researchers nor the participants know what treatment the subjects is receiving), randomized, placebo-controlled. It consists of 3 phases: a Screening phase, a Treatment phase and a Follow-up phase. In Treatment phase participants will be randomly assigned VX-787, 600 mg or placebo 2 times a day, on Day 1 to 9, followed by a single dose of VX-787 600 mg or placebo in the morning on Day 10. Pharmacokinetic parameters will be assessed primarily. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Female participants must be of non-childbearing potential: postmenopausal for at least 2 years (amenorrheal for at least 3 years and a serum follicle stimulating hormone [FSH] level greater than [>] 40 international unit per liter [IU/L]), or surgically sterile (have had a total hysterectomy, bilateral oophorectomy, or bilateral tubal ligation/bilateral tubal clips without reversal operation), or otherwise incapable of becoming pregnant
* Participants must be non-smoking or smoking no more than 10 cigarettes, or 2 cigars, or 2 pipes per day for at least 3 months prior to screening
* Participants must have a Body Mass Index (BMI: weight in kg divided by the square of height in meters) of 18.0 to 30.0 kilogram per meter square [kg/m^2]
* Participants must be willing/able to adhere to the prohibitions and restrictions specified in the protocol and study procedures
* Participants must be healthy on the basis of a medical evaluation that reveals the absence of any clinically significant abnormality and includes a physical examination, medical history, vital signs and the results of blood biochemistry, blood coagulation and hematology test and a urinalysis performed at screening

Exclusion Criteria:

* Participants with a past history of heart arrhythmias (for example, extrasystoli, tachycardia at rest), history of risk factors for Torsade de Pointes syndrome (for example, hypokalemia, family history of long QT Syndrome)
* Participants with a history or evidence of use of alcohol, barbiturates, amphetamines, recreational or narcotic drug use within the past 1 year, which in the Investigator's opinion would compromise participant's safety and/or compliance with the study procedures
* Participants with current hepatitis A infection (confirmed by hepatitis A antibody immunoglobulin M [IgM]), or hepatitis B infection (confirmed by hepatitis B surface antigen [HBsAg]), or hepatitis C infection (confirmed by hepatitis C virus [HCV] antibody), or human immunodeficiency virus type 1 (HIV-1) or HIV-2 infection at study screening
* Participants having a positive urine drug test or alcohol breath test at study screening. Urine will be tested for the presence of amphetamines, benzodiazepines, cocaine, cannabinoids, opioids, methadone and barbiturates
* Participants with known allergies, hypersensitivity, or intolerance to VX-787, oseltamivir, or excipients of the drug products used

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Assess the drug-drug interaction between VX-787 600 mg bid coadministered with oseltamivir 75 mg bid at steady-state in healthy participants | Day 5
  Based on the individual plasma concentration-time data, using the actual sampling times the following PK parameters will be derived: Ctrough, Cmin, Cmax, tmax, AUC12h, Cavg, FI Ratio Cmax,test/refrence (ref), Ratio Cmin,test/ref and ratio AUC12h, test/ref
Evaluate the safety and tolerability of a VX-787 600 mg bid regimen during 10 days in healthy participants | Days 1-10
  Safety and tolerability will be evaluated throughout the study from signing of the ICF onwards until the last study-related activity. The study will include the following evaluations of safety and tolerability: Adverse Events, Clinical Laboratory Test, Electrocardiograms, Vital Signs, Physical Exams.
Assessment of Pharmacokinetics of VX-787 | Days 1-10
  Pharmacokinetic parameters will include assessment of Ctrough, Cmin, Cmax, tmax, AUC12h, Cavg, FI Ratio Cmax,test/ref, ratio Cmin,test/ref and ratio AUC12h,test/ref.

SECONDARY OUTCOMES:
Investigate the short-term safety and tolerability of the concomitant use of VX-787 and oseltamivir in healthy participants | Days 1-5
  Safety and tolerability will be evaluated throughout the study from signing of the ICF onwards until the last study-related activity. The study will include the following evaluations of safety and tolerability: Adverse Events, Clinical Laboratory Test, Electrocardiograms, Vital Signs, Physical Exams

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Infectious Diseases BVBA Clinical Trial, Study Director — Janssen Infectious Diseases BVBA
Locations (1):
- Merksem, Belgium